CLINICAL TRIAL: NCT01176604
Title: A Humanitarian Device Exemption Treatment Protocol of TheraSphere® for Treatment of Unresectable Hepatocellular Carcinoma
Brief Title: Yttrium Y 90 Glass Microspheres in Treating Patients With Unresectable Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0770; NCI-2018-01816 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2008-0770 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2010-08-04; First posted 2010-08-06 (Estimated); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Stage III Hepatocellular Carcinoma AJCC v8; Stage IIIA Hepatocellular Carcinoma AJCC v8; Stage IIIB Hepatocellular Carcinoma AJCC v8; Stage IV Hepatocellular Carcinoma AJCC v8; Stage IVA Hepatocellular Carcinoma AJCC v8; Stage IVB Hepatocellular Carcinoma AJCC v8; Unresectable Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (yttrium Y 90 glass microspheres) (Experimental): Patients receive yttrium Y 90 glass microspheres via a catheter over 5 minutes on day 0. Patients may receive additional treatments at 4-12 week intervals until all tumors in the liver have been treated in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Yttrium Y 90 Glass Microspheres

INTERVENTIONS:
Radiation: Yttrium Y 90 Glass Microspheres — Given via catheter
  Other Names: TheraSphere

SUMMARY:
This trial studies how well yttrium Y 90 glass microspheres work in treating patients with hepatocellular carcinoma that cannot be removed by surgery. Radioactive drugs, such as yttrium Y 90 glass microspheres, may carry radiation directly to cancer cells and not harm normal cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Provide oversight to treatment with yttrium Y 90 glass microspheres (TheraSphere) to eligible patients with hepatocellular carcinoma (HCC) of the liver who are not surgical resection candidates.

II. Evaluate patient experience, toxicities and overall survival associated with TheraSphere treatment.

OUTLINE:

Patients receive yttrium Y 90 glass microspheres via a catheter over 5 minutes on day 0. Patients may receive additional treatments at 4-12 week intervals until all tumors in the liver have been treated in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 3-6 weeks, then annually for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of intrahepatic HCC. The histopathology confirmation criterion may be waived in patients with a radiographically identifiable liver mass, known laboratory or clinical risk factors for cancer or elevated tumor markers such as alphafetoprotein (AFP) and clinical findings. Guidelines from the American Association for the Study of Liver Diseases (AASLD) and the European Association for the Study of the Liver (EASL) describe in detail the approach and algorithm for diagnosing HCC
* Eastern Cooperative Oncology Group (ECOG) Performance Status Score 0 - 2
* Life expectancy >= 3 months
* > 4 weeks since prior radiation, surgery or chemotherapy
* Able to comprehend and provide written informed consent in accordance with institutional and federal guidelines

Exclusion Criteria:

* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 5 times upper normal limit (UNL) (within 15 days of treatment demonstrating liver dysfunction)
* Serum bilirubin > 2.0 mg/dl (unless segmental infusion is planned) (within 15 days of treatment demonstrating liver dysfunction)
* Any contraindications to angiography and hepatic artery catheterization such as:

  * History of severe allergy or intolerance to any contrast media, narcotics, sedatives, or atropine that cannot be corrected or premedicated
  * Bleeding diathesis, not correctable by usual forms of therapy
  * Severe peripheral vascular disease that would preclude catheterization
* Evidence of potential delivery of greater than 16.5 mCi (30 Gy absorbed dose) of radiation to the lungs in a single treatment
* Clinical evidence of pulmonary insufficiency
* Evidence of any detectable technetium-99 macroaggregated albumin (Tc-99m MAA) flow to the stomach or duodenum, after application of established angiographic techniques to stop or mitigate such flow
* Complete occlusion of the main portal vein
* Significant extrahepatic disease representing an imminent life-threatening outcome
* Active uncontrolled infection
* Significant underlying medical or psychiatric illness
* Co-morbid disease of condition that would preclude safe delivery of TheraSphere treatment or, in the judgment of the physician, place the patient at undue risk
* Pregnancy
* Tumor type demonstrated on imaging to be infiltrative, tumor volume > 70% of the target liver volume, or tumor nodules too numerous to count, or tumor volume > 50% combined with an albumin < 3 g/dL, or complete occlusion of the main portal vein

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2010-08-04 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
Oversight to treatment with yttrium Y 90 glass microspheres | Up to 2 years
  Associated with yttrium Y 90 glass microspheres treatment. Data analysis will be limited to descriptive reports of the number and characteristics of the patients treated and their clinical and adverse event experiences.
Patient experience | Up to 2 years
  Associated with yttrium Y 90 glass microspheres treatment. Data analysis will be limited to descriptive reports of the number and characteristics of the patients treated and their clinical and adverse event experiences.
Incidence of adverse events | 30 days after each treatment
  Associated with yttrium Y 90 glass microspheres treatment. Data analysis will be limited to descriptive reports of the number and characteristics of the patients treated and their clinical and adverse event experiences.
Overall survival | Up to 2 years
  Associated with yttrium Y 90 glass microspheres treatment. Data analysis will be limited to descriptive reports of the number and characteristics of the patients treated and their clinical and adverse event experiences.

CONTACTS AND LOCATIONS:
Overall Officials: Armeen Mahvash, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org